CLINICAL TRIAL: NCT07008378
Title: A Phase I, Multicenter, Open-Label Study to Evaluate the Safety, Tolerability, Cellular Kinetics, and Pharmacodynamics of P-CD19CD20-ALLO1 in Patients With Multiple Sclerosis
Brief Title: A Study to Evaluate the Safety, Tolerability, Cellular Kinetics, and Pharmacodynamics of P-CD19CD20-ALLO1 in Participants With Multiple Sclerosis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Genentech, Inc. (Industry)
Collaborators: Poseida Therapeutics, Inc., a member of the Roche Group (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GN45773
Record Dates: First submitted 2025-05-20; First posted 2025-06-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Dose Escalation (Experimental): Participants will receive a lymphodepleting chemotherapy regimen followed by a single infusion of P-CD19CD20-ALLO1. Dose escalation decisions will be made after participants are observed for a minimum of 28 days for toxicity.
  Interventions: Biological: P-CD19CD20-ALLO1 Cells; Drug: Cyclophosphamide; Drug: Fludarabine

INTERVENTIONS:
Biological: P-CD19CD20-ALLO1 Cells — P-CD19CD20-ALLO1 Cells will be administered intravenously as per the schedule specified in the protocol.
Drug: Cyclophosphamide — Cyclophosphamide will be administered intravenously.
Drug: Fludarabine — Fludarabine will be administered intravenously.

SUMMARY:
This study aims to explore the safety, tolerability, cellular kinetics, and pharmacodynamics of P-CD19CD20-ALLO1 in participants with progressive multiple sclerosis (PMS) and relapsing multiple sclerosis (RMS).

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years (inclusive) at the time of signing Informed Consent Form
* Diagnosis of progressive MS according to the revised McDonald 2017 criteria, and:

Expanded disability status scale (EDSS) score at screening, from 3 to 6 inclusive Evidence of disability progression and no relapses in the 2 years prior to screening

- Diagnosis of relapsing MS according to the revised McDonald 2017 criteria, and: Evidence of clinical relapses and MRI activity within two years prior to screening while on a disease modifying therapy

* EDSS score at screening, from 0 to 6 inclusive
* No relapses within 45 days of screening

Exclusion Criteria:

* Pregnant or breastfeeding, or intention of becoming pregnant within the timeframe in which contraception is required
* Participants who have confirmed or suspected Progressive Multifocal Leukoencephalopathy (PML)
* Known or suspected history of Hemophagocytic Lymphohistiocytosis/ Macrophage Activation Syndrome (HLH/MAS) or neurotoxicity with prior therapies
* Known presence of other neurologic disorders that may mimic MS
* History of currently active primary or secondary (non-drug-related) immunodeficiency
* Significant or uncontrolled medical disease which would preclude patient participation
* High risk for clinically significant bleeding or any condition requiring plasmapheresis, IV Ig, or acute blood product transfusions
* History of recurrent serious infections or chronic infection
* Prior treatment with CAR T-cell therapy, gene-therapy product, total body irradiation, bone marrow transplantation, allograft organ transplant, or hematopoietic stem cell transplant at any point
* Any previous treatment with immunomodulatory or immunosuppressive medication without an appropriate washout period.
* Inability to complete an MRI scan

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-15 (Actual); Primary Completion 2032-08-31 (Estimated); Study Completion 2032-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Dose-limiting Toxicity (DLTs) at Each Dose Level of P-CD19CD20-ALLO1 | Day 1 up to Day 29
Number of Participants With Adverse Events (AEs) | Up to 5 years

SECONDARY OUTCOMES:
Number of Chimeric Antigen Receptor (CAR) Transgene Copies in Blood Assessed by Droplet Digital Polymerase Chain Reaction (ddPCR) | Up to 5 years
B-cell Levels in the Blood | Up to 5 years
Number of Participants With Anti-CAR T Antibodies | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Genentech, Inc.
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No